CLINICAL TRIAL: NCT00389636
Title: TheraGauze™ Alone and Regranex®Gel 0.01% Plus TheraGauze™ in the Treatment of Wagner Stage I Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Solsys Medical LLC (Industry)
Responsible Party: Allan Staley, Soluble Systems, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SS-0601
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes; Foot; Extremity; Ulcer; Wound; Gauze
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Ulcer; Wounds and Injuries | interventions — Becaplermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): TheraGauze alone
  Interventions: Device: TheraGauze
- 2 (Active Comparator): Theragauze + Regranex
  Interventions: Drug: Regranex

INTERVENTIONS:
Device: TheraGauze — TheraGauze
  Arms: 1
Drug: Regranex — Regranex + TheraGauze
  Arms: 2

SUMMARY:
Patients will be randomized to receive TheraGauze alone or with Regranex to treat diabetic foot ulcer condition. The purpose of the study is provide the sponsor with pilot information regarding the ability of TheraGauze to promote wound healing on its own and to examine synergy with Regranex in the treatment of diabetic foot ulcers.

DETAILED DESCRIPTION:
This study will evaluate the use of TheraGauzeT (Soluble Systems, LLC) wound dressing, a polymer hydrogel chemically impregnated into a rayon/polyester formed fabric, forming a pliable, conforming solid matrix. TheraGauze is FDA Class I exempt (regulation #21CFR, product code 5878.4022). It is hypothesized that this material will be useful for the treatment of full-thickness diabetic ulcers. It is further hypothesized that this material will enhance the action of Regranex (becaplermin) gel by providing an optimal environment for this growth factor to function. This study will observe patient outcomes following diabetic foot ulcer treatment with TheraGauze and with or without the use of Regranex.

ELIGIBILITY:
Inclusion Criteria: Patients

* who are 18 years old or older;
* who are diagnosed as having insulin-dependent or non-insulin-dependent diabetes mellitus (5.5% <HgBA1C<12%);
* who have foot ulcers extending through the epidermis and dermis but not with exposed tendon or bone;
* who have a diagnosis of chronic diabetic ulcer;
* who have a viable wound bed with granulation tissue as determined by bleeding following debridement;
* who have an ulcer size which is at least 1 cm2 and no greater then 16cm2;
* who have signed an informed consent form.
* who have a wound that has been present for at least 4 weeks at the time of screening.

Exclusion Criteria: Patients

* having ulcers less than 1cm2 or greater than 16cm2 in size;
* having severe arterial disease (ankle brachial index (ABI) less than 0.65);
* having history of radiation therapy to the ulcer site;
* who use corticosteroids >10mg prednisone daily
* who use any immune suppressive, or severely immunocompromised patients;
* who have an ulcer that was of a non-diabetic pathophysiology;
* having vasculitis, severe rheumatoid arthritis, or other collagen vascular disease;
* having malnutrition (defined by albumin <2.5 g/dL);
* having a known allergy or hypersensitivity to the components of either TheraGauze or Regranex;
* having erythema or purulence associated with a severe infection of the wound site;
* having signs and symptoms of cellulitis, osteomyelitis, necrotic or avascular ulcer beds;
* undergoing hemodialysis;
* having uncontrolled diabetes (defined as HgB A1c>12%)
* having deficient blood supply to ulcers (defined as capillary fill time >3 seconds at tips of toes)
* having Charcot's neuroarthropathy as determined by clinical and/or radiographic examination;
* having sickle cell disease;
* having exposed bone, tendon, or fascia;
* who are currently enrolled in a clinical evaluation of another investigational device or drug, or have received and investigational treatment for diabetic foot ulcers in the last 30 days;
* unable to comply with the procedures described in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-09; Primary Completion 2008-07 (Estimated); Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Frequency of complete wound healing within 12 weeks
Time to complete wound healing within 12 weeks

SECONDARY OUTCOMES:
Investigator's or clinician's assessment of wound quality (ulcer duration, baseline area, staging, presence of fibrin or granulation tissue)
Patient's assessment (pain, itching)
Presence of epithelialization visible on the wound surface
Occurrence of infection at the wound site
Recurrence of ulcer during the 20 week follow-up period
Adverse events (infection, cellulites, seroma, etc.)
Excess pain

CONTACTS AND LOCATIONS:
Overall Officials: Anne Laumann, MBChB, MRCP, Principal Investigator — Northwestern University; Adam Landsman, DPM, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States